CLINICAL TRIAL: NCT04712292
Title: Effects of the COVID-19 Pandemic on the Diagnosis, Treatment and Outcomes of Patients Affected by Colorectal Cancer Requiring Surgery: Results From a National Multicentre Cohort Study
Brief Title: Effects of COVID-19 Pandemic on the Outcomes of Colorectal Cancer
Acronym: COVID-CRC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Matteo Rottoli, Professor, University of Bologna
Other Study IDs: 854/2020/Oss/AOUBo
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Colorectal Neoplasms Malignant
Keywords: colorectal cancer; diagnosis; screening; COVID-19; surgery; outcomes
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Disease; COVID-19 | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Patients undergoing surgery for confirmed or suspected colorectal cancer between January 2020 and December 2021
  Interventions: Procedure: Surgical procedure for confirmed or suspected colorectal cancer
- Control group: Patients undergoing surgery for confirmed or suspected colorectal cancer between January 2018 and December 2019
  Interventions: Procedure: Surgical procedure for confirmed or suspected colorectal cancer

INTERVENTIONS:
Procedure: Surgical procedure for confirmed or suspected colorectal cancer — Surgical procedure for cancer may include:
  * any radical surgery (right or left hemicolectomy, rectal resection, abdomino-perineal resection, total colectomy, proctocolectomy, and others depending on the tumor site and other tumor characteristics),
  * surgery for radicalization of cancer polyps previously removed endoscopically
  * surgery for excision of large polyps which are not removable endoscopically
  * staging surgery (laparoscopy or laparotomy), in case of advanced-non operable cancer
  * palliative surgery (defined as any surgery with no curative intent)

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection has been identified as the cause of the Coronavirus disease 19 (COVID-19), which was initially reported in December 2019 in China and has since rapidly spread worldwide.

Since then, the COVID-19 pandemic has caused a detrimental effect of the national health care system, causing a drastic reduction of the screening programs for colorectal cancer and requiring the redistribution of the hospital resources from elective surgery to the care of patients with SARS-Cov_2 infection requiring admission.

DETAILED DESCRIPTION:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection has been identified as the cause of the Coronavirus disease 19 (COVID-19), which was initially reported in December 2019 in China and has since rapidly spread worldwide. Italy witnessed a rapid and uncontrolled spread of the infection after March 2020, and a worrisome increasing number of related deaths.

The need for increased capacity for COVID-19 patients required elective activities to be drastically reduced or canceled. The unprecedented stress on the healthcare system has caused the reduction of the elective surgery and the cancer screening programs during the last 2 years. Studies predicting harmful impact of the COVID-19 pandemic on cancer care have been already published. However, it has not been proved whether the potential delay of screening, diagnosis and treatment could have a measurable effect on patients undergoing surgery for colorectal cancer in the COVID-19 era.

The aim of the study is therefore to compare the 30-day perioperative and oncologic outcomes between patients undergoing surgery for cancer of the colon and rectum between January 2020 and December 2021 (study group) and those who had surgery for colorectal cancer between January 2018 and December 2019 (Control Group), in order to identify:

* any change in the distribution of the histological stage (primary aim)
* any change in the rate of palliative surgery (primary aim)
* any change in the rate of non-radical surgery (R1 or R2 resection) ( primary aim)
* any change in the rate of 30-day postoperative complications (secondary outcome)

Anonimyzed data will be retrospectively collected on a RedCap platform hosted on the servers of the Alma Mater Studiorum University of Bologna. The variables included demographic characteristics, comorbidities, details of the disease at the diagnosis, details of the neoadjuvant therapy, perioperative variables and 30-day postoperative follow-up variables.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing radical surgery for histologically confirmed diagnosis of cancer located in the colon, the rectum or the anus; or
* any patient undergoing surgery with oncologic intents, for instance: radicalization of endoscopically removed cancerous polyp; radical surgery to remove large, at-risk polyp which are not removable by endoscopy; or
* any patient undergoing planned or unpredicted palliative surgery for a primary cancer localized in the colon, rectum or anus; or
* any patient undergoing a staging procedure (i.e. staging laparoscopy, surgical exploration), which did not result in any radical surgery due to advanced disease, metastasis, etc.

and

* age > 18 years
* elective or urgent surgery

Exclusion Criteria:

* Colorectal cancer recurring after previous surgery;
* Cancer originating from other organs than the colon, the rectum and the anus;
* Lack of significant histological details (expect when the cancer was not removed)
* lack of 30-day follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include all adult patients undergoing elective or urgent surgery for proven or suspected colorectal within the study periods
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2022-02-15 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Oncologic stage | 30 days from the surgery
  The stage will be reported at the histological examination according to TNM classification
Palliative surgery | at time 0 (surgery)
  Rate of palliative surgery (defined as any procedure which did not have the aim of radically removing the primary cancer, either planned preoperatively in order to reduce the symptoms, or which became necessary during surgery due to unexpected findings
Rate of radical surgery | 30 days from surgery
  Surgery is defined radical according to the absence of cancer (R0) at the surgical margins on the histological specimen

SECONDARY OUTCOMES:
Aggressive cancer biology | 30 days from the surgery
  Biology was considered aggressive if any of the following characteristics were found at the histological examination: signet ring cells, mucinous tumor, tumor budding, lymphovascular invasion, perineurial invasion, lymphangitis.
Rate of clinical T4 cancer at the preoperative staging | At time 0 (surgery)
  Clinical T4 cancer are defined as those with high suspicious of local invasion of adjacent organs or structures, not necessary confirmed as T4 at the histological examination
Liver metastases | At the preoperative staging or at surgery (time 0)
  Rate of single/multiple liver metastases
Lung metastases | At the preoperative staging or at surgery (time 0)
  Rate of single/multiple lung metastases
Associated symptoms | Before surgery
  Rate of patients who had a diagnosis of cancer without any associated symptoms - as sign of effectiveness of the screening
Emergency surgery | surgery (time 0)
  rate of operations requiring surgery within 48 hours from the unpredicted admission to hospital
Postoperative complications | 30 days from surgery
  Rate of 30-day complications graded according to the Clavien-Dindo Classification
Mortality | 30 days from surgery
  Rate of 30-day deaths

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Rottoli, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna, Alma Mater Studiorum University of Bologna
Locations (44):
- Italy (44):
  - Rho Memorial Hospital, Rho, Milan
  - Humanitas Research Center, Rozzano, Milan
  - AOU Policlinico di Bari "M. Rubino", Bari
  - Policlinico di Bari, Bari
  - Humanitas Gavazzeni Hospital, Bergamo
  - Policlinico San Marco, Bergamo
  - Maggiore Hospital, Bologna
  - Fondazione Poliambulanza, Brescia
  - Spedali Civili, Brescia
  - Santissima Trinità Hospital, Cagliari
  - Vittorio Emanuele III Hospital, Carate Brianza
  - San Paolo Hospital, Civitavecchia
  - AUSL Romagna Ravenna-Faenza, Faenza
  - San Giovanni di Dio Hospital, Florence
  - Gardone Val Trompia Hospital, Gardone Val Trompia
  - ASST FBF Sacco Hospital, Milan
  - San Raffaele Hospital, Milan
  - ASST Santi Paolo e Carlo Hospital, Milan
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico - Milano, Milan
  - Istituto Nazionale dei Tumori, Milan
  - Mirano Hospital, Mirano
  - AORN Cardarelli, Napoli
  - Università della Campania Luigi Vanvitelli, Napoli
  - Padova University Hospital, Padua
  - Veneto Institute of Oncology IOV-IRCCS, Padua
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia-Cervello, Palermo
  - AOU Parma, Parma
  - San Matteo Hospital, Pavia
  - Pederzoli Hospital, Peschiera del Garda
  - Azienda Sanitaria Fiuli Occidentale, Pordenone
  - Ceccarini Hospital, Riccione
  - Infermi Hospital, Rimini
  - Campus Biomedico, Roma
  - Fondazione Policlinico Roma Tor Vergata, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - San Filippo Neri Hospital, Roma
  - Sant'Eugenio Hospital, Roma
  - UOSD Tor Vergata, Roma
  - AOU Sassari, Sassari
  - Regional Hospital Treviso, Treviso
  - University Hospital of Trieste, Trieste
  - AOU Città della Salute e della Scienza, Turin
  - Mauriziano Hospital, Turin
  - ASST Vimercate, Vimercate

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Greenwood E, Swanton C. Consequences of COVID-19 for cancer care - a CRUK perspective. Nat Rev Clin Oncol. 2021 Jan;18(1):3-4. doi: 10.1038/s41571-020-00446-0. PMID 33097915
- [Result] Jazieh AR, Akbulut H, Curigliano G, Rogado A, Alsharm AA, Razis ED, Mula-Hussain L, Errihani H, Khattak A, De Guzman RB, Mathias C, Alkaiyat MOF, Jradi H, Rolfo C; International Research Network on COVID-19 Impact on Cancer Care. Impact of the COVID-19 Pandemic on Cancer Care: A Global Collaborative Study. JCO Glob Oncol. 2020 Sep;6:1428-1438. doi: 10.1200/GO.20.00351. PMID 32986516
- [Result] Torzilli G, Vigano L, Galvanin J, Castoro C, Quagliuolo V, Spinelli A, Zerbi A, Donadon M, Montorsi M; COVID-SURGE-ITA group. A Snapshot of Elective Oncological Surgery in Italy During COVID-19 Emergency: Pearls, Pitfalls, and Perspectives. Ann Surg. 2020 Aug;272(2):e112-e117. doi: 10.1097/SLA.0000000000004081. PMID 32675512
- [Result] Mitchell EP. Declines in Cancer Screening During COVID-19 Pandemic. J Natl Med Assoc. 2020 Dec;112(6):563-564. doi: 10.1016/j.jnma.2020.12.004. No abstract available. PMID 33339569
- [Result] Onder G, Rezza G, Brusaferro S. Case-Fatality Rate and Characteristics of Patients Dying in Relation to COVID-19 in Italy. JAMA. 2020 May 12;323(18):1775-1776. doi: 10.1001/jama.2020.4683. No abstract available. PMID 32203977